CLINICAL TRIAL: NCT01736592
Title: An Open Label Study to Determine the Long Term Safety, Tolerability and Biological Activity of SAR422459 in Patients With Stargardt's Macular Degeneration
Brief Title: Phase I/II Follow-up Study of SAR422459 in Patients With Stargardt's Macular Degeneration
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LTS13588; SG1/002/11 (Other: Sanofi Identifier); 2024-513501-31 (Registry Identifier: CTIS); 2012-001990-95 (EudraCT Number)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stargardt's Disease
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Long Term Follow up (Other): Long term follow up in all patients who received SAR422459 in previous study TDU13583
  Interventions: Drug: Long term follow up in all patients who received SAR422459 in previous study TDU13583

INTERVENTIONS:
Drug: Long term follow up in all patients who received SAR422459 in previous study TDU13583 — Blood draw for the laboratory assessment

SUMMARY:
Primary Objective:

To evaluate the long-term safety and tolerability of SAR422459 in patients with Stargardt's Macular Degeneration.

Secondary Objective:

To assess:

* Safety
* Biological activity

DETAILED DESCRIPTION:
Patients will be followed for 15 years after completion/early termination from the previous TDU13583 study (NCT01367444).

As the initial TDU13583 study is terminated - recruitment to this LTS13588 study is over with 27 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria:

1. Provide signed and dated written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA])
2. Must have been enrolled in protocol TDU13583 (SG1/001/10)
3. Must have received a subretinal injection of SAR422459
4. Must have completed protocol TDU13583 to Week 48 or undergone an early discontinuation visit.

Exclusion Criteria:

The following would exclude Patients from participation in the study:

1. Did not receive SAR422459 as part of the TDU13583 protocol.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2033-08-29 (Estimated); Study Completion 2033-08-29 (Estimated)

PRIMARY OUTCOMES:
The incidence of Adverse Events | 15 years
  The number and percentage of patients with treatment emergent adverse events

SECONDARY OUTCOMES:
Clinically important changes in ocular safety assessments | baseline to 15 years
  From baseline in (TDU13583) study and from the last visit best-corrected visual acuity (BCVA), slit-lamp examination, Fundososcopy, intraocular pressure, laboratory parameters, concomitant medications
Delay in retinal degeneration | baseline to 15 years
  Measured as change from baseline in function relative to untreated contralateral eye on: BCVA, static perimetry, microperimetry, autofluorescence, optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (2):
- Oregon Health and Science University Site Number : 840001, Portland, Oregon, United States
- Investigational Site Number : 250001, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org